CLINICAL TRIAL: NCT06452563
Title: Amino Acids Supplementation and Exercise Intervention in Hemodialysis Patients: Effects on Muscle and Fatigue - a Randomized Controlled Trial
Brief Title: Amino Acids Supplementation and Exercise Intervention in Hemodialysis Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Emad Magdy, Associate Professor Of Nephrology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.24.04.2576
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis Complication; Malnutrition
Keywords: haemodialysis patients; ketoanalogs; malnutrition; exercise; Muscle function
MeSH Terms: conditions — Malnutrition; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketoanalogs Supplementation Group (Active Comparator): Participants will receive daily a total of six tablets of Ketoanalogs Supplementation divided into three doses for three months .
  Interventions: Dietary Supplement: ketoanalogue supplementation
- Ketoanalogs Supplementation and intradialytic exercise group (Active Comparator): Participants will receive daily a total of six tablets of Ketoanalogs Supplementation divided into three doses for three months in addition to doing intradialytic exercise .
  Interventions: Dietary Supplement: ketoanalogue supplementation; Other: intradialytic exercise
- Intradialytic exercise group (Active Comparator): Participants will be asked to do intradialytic exercise only
  Interventions: Other: intradialytic exercise
- Control group (No Intervention): Participants will not receive drug or do exercises

INTERVENTIONS:
Dietary Supplement: ketoanalogue supplementation — This drug contains 5 essential amino acids (L-lysine monoacetate 75mg, L-threonine 53mg, L-tryptophan 23mg, L-histidine 38mg and L-tyrosine 30mg) and 5 essential amino acid substitutes in the form of calcium salts, including 4 keto-analogues (keto-isoleucine, keto-leucine, keto-valine, and keto-phenylalanine) and a hydroxy-analogue (hydro methionine) as calcium salt . The drug is approved by the Egyptian Drug Authority (EDA) with registration number 34677/2021
  Arms: Ketoanalogs Supplementation Group; Ketoanalogs Supplementation and intradialytic exercise group
Other: intradialytic exercise — low-intensity exercise training composed of knee extension and hip abduction and flexion from a three-repetition maximum (3RM) using ankle weights
  Arms: Intradialytic exercise group; Ketoanalogs Supplementation and intradialytic exercise group

SUMMARY:
The goal of this randomized clinical trial is to observe the effect of Amino acids (AAs)supplementation and exercises in haemodialysis patients . The main question it aims to answer is :

Does AAs supplementation and regular exercises have an effect on the muscle mass and function in haemodialysis patients ? Participants will receive daily a total of six tablets of amino acids supplementation divided into three doses. And some Participants will also be asked to do intradialytic exercise.

Researchers will compare the effects of these interventions on the muscle mass and fatigue, among four groups:

1. A group that will be only taking AAs supplementation
2. A group taking AAs supplementation along with intradialytic exercise
3. A group only performing intradialytic exercise
4. A passive control group This will be monitored through BMI, anthropometric measures, Musculoskeletal ultrasound assessment of the quadriceps muscle , fatigue questionnaires and sit and stand test.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients due to chronic kidney diseases
* Age between 18 - 60

Exclusion Criteria:

* Frail patients
* The patients who refused to participate
* Growth retarded patients
* Disabilities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 3 months
  skeletal muscle mass (SMM) will be assessed using the Inbody test before and after this trial .
Muscle function test | 3 months
  The muscle function will be assessed by the Sit-to-Stand Test (STS) . The test is comprised of counting the maximum number of times that the subject is able to stand up unassisted or assisted from a chair in 30 seconds .
The thickness of the quadriceps rectus femoris and quadriceps vastus intermedius | 3 months
  The thickness of the quadriceps rectus femoris (QRFT) and quadriceps vastus intermedius (QVIT) will be assessed before and after this trial using Ultrasonography. The measurements will be conducted in a standardized manner at two specific landmarks: the midpoint and the border between the lower third and upper two-thirds between the superior anterior iliac spine and the upper pole of the patella .

SECONDARY OUTCOMES:
Fatigue score | 3 months
  Fatigue score will be measured pre- and post- this trial using the Modified Fatigue Impact Scale (MFIS) . Higher MFIS scores indicate a higher burden of fatigue, and less physical activity, concentration, or motivation, respectively. A subjective fatigue score of ≥35 was defined as severe fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No